CLINICAL TRIAL: NCT06339905
Title: Evaluation of the Effects of EndoActivator Use on Postoperative Pain and Root Canal Treatment Success
Brief Title: The Effects of EndoActivator on Postoperative Pain and Root Canal Treatment Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, yeldaerdem, Director, Clinical Research, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-772.02-5564
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Periapical Periodontitis; Root Canal Infection
Keywords: Chronic apical periodontitis; irrigation activation; periapical index; postoperative pain; treatment outcome; periapical health
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonic Activation with EndoActivator (Experimental): Sonic irrigation was performed using an EndoActivator sonic handpiece (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA). A suitable-size activator tip was selected and loosely placed at 2 mm from working length, and the device was operated at 10,000 cycles/min using a pumping action to move the tip to produce vertical strokes of 2-3 mm.
  Interventions: Procedure: Sonic Activation with EndoActivator
- Conventional needle irrigation (control) (Active Comparator): Conventional needle irrigation was performed with short, in-and-out vertical strokes of 2-3 mm at a rate of approximately 100 strokes per minute.
  Interventions: Procedure: Control Needle Irrigation

INTERVENTIONS:
Procedure: Sonic Activation with EndoActivator — sonic activation
  Other Names: EndoActivator (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA)
  Arms: Sonic Activation with EndoActivator
Procedure: Control Needle Irrigation — control group
  Other Names: CNI
  Arms: Conventional needle irrigation (control)

SUMMARY:
This study evaluates postoperative pain and radiographic healing of asymptomatic posterior teeth with chronic apical periodontitis following root-canal treatment performed using EndoActivator for irrigation activation.

DETAILED DESCRIPTION:
Aim: To evaluate postoperative pain and radiographic healing of asymptomatic posterior teeth with chronic apical periodontitis following root-canal treatment performed using EndoActivator for irrigation activation.

Methodology: In this clinical trial, root-canal treatment was performed on 140 posterior teeth with chronic apical periodontitis. After routine canal preparation, patients were assigned to either a control group treated using conventional needle irrigation (CNI) without activation or to sonic irrigation activation with EndoActivator. All treatment was completed in a single visit. Patients provided self-assessments of the severity of postoperative pain at 1, 2,3 and 7 days using a Verbal Rating Scale (VRS) and Wong Baker Face Scale. Patients were recalled at 12 months for clinical and radiographic examinations. Periapical healing was evaluated using a periapical index (PAI), with scores of 1 or 2 considered to represent treatment success and scores of 3, 4, or 5 to represent treatment failure. Data were analyzed using one-way ANOVA and Kruskal-Wallis tests, with differences of P < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 patient's age
* Being systemically healthy
* Having posterior teeth (molar or premolar) with chronic apical periodontitis lesion (PAI≥3)

Exclusion Criteria:

* Clinically symptomatic teeth
* Patients with complicated systemic disease (ASA 3 - 6)
* Teeth with open apex
* Teeth having curvature more than 20 degree
* Not having enough tooth structure to be isolated with rubber dam
* Patients with severe periodontal defects or deep periodontal pockets (probing depth> 4 mm)
* A history of taking analgesics 12 hours ago or antibiotics 1 month ago
* Patients who cannot come to control sessions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
change from baseline postoperative pain at 1 week | 1,2,3 and 7 days
  Pain was measured using a Verbal Rating Scale with 4 levels, as follows: 0, no pain; 1, slight pain (mild discomfort, no treatment needed); 2, moderate pain (pain required analgesics for relief); 3, severe pain (pain and/or swelling not relieved by simple analgesics and required unscheduled visit) and Wong Baker Face Scale with six different facial expression. Patients were provided forms and asked to record preoperative pain as well as pain at 1,2,3 and 7 days postoperatively, and to note down the number of analgesics taken. Patients returned their completed forms at their 1-week follow-up visits.
change from baseline periapical index at 1 year | Clinical and radiographic examinations were performed on the 1 day of treatment, and 1 year after treatment.]
  Periapical tissue was evaluated using a 5-point periapical index (PAI) (Ørstavik et al. 1986) and scored as follows: 1: Normal periapical structures; 2: Small changes in bone structures; 3: Changes in bone structure with some mineral loss; 4: Periodontitis with well-defined radiolucent area; 5: Severe periodontitis with exacerbating features.
  Treatment was considered successful if the patient had no discomfort, no percussion/palpation pain, no sinus tract, no mobility or associated soft-tissue swelling, and a PAI score of ≤ 2. Treatment was considered a failure if the patient could not perform normal masticatory functions, experienced discomfort and percussive pain upon examination, and/or had a PAI score of ≥ 3 .

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Ersahan, PhD, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After its publication in a journal, the investigators want to share their data.
Supporting Information: Study Protocol, SAP
Time Frame: After its publication in a journal, the investigators want to share their data.
Access Criteria: Postoperative pain scores, radiographic and clinical findings.

REFERENCES:
- [Background] Orstavik D. Time-course and risk analyses of the development and healing of chronic apical periodontitis in man. Int Endod J. 1996 May;29(3):150-5. doi: 10.1111/j.1365-2591.1996.tb01361.x. PMID 9206419
- [Background] Ramamoorthi S, Nivedhitha MS, Divyanand MJ. Comparative evaluation of postoperative pain after using endodontic needle and EndoActivator during root canal irrigation: A randomised controlled trial. Aust Endod J. 2015 Aug;41(2):78-87. doi: 10.1111/aej.12076. Epub 2014 Sep 4. PMID 25195661
- [Background] Swimberghe RCD, Buyse R, Meire MA, De Moor RJG. Efficacy of different irrigation technique in simulated curved root canals. Lasers Med Sci. 2021 Aug;36(6):1317-1322. doi: 10.1007/s10103-021-03263-8. Epub 2021 Feb 23. PMID 33624186
- [Background] Brito PR, Souza LC, Machado de Oliveira JC, Alves FR, De-Deus G, Lopes HP, Siqueira JF Jr. Comparison of the effectiveness of three irrigation techniques in reducing intracanal Enterococcus faecalis populations: an in vitro study. J Endod. 2009 Oct;35(10):1422-7. doi: 10.1016/j.joen.2009.07.001. PMID 19801244